CLINICAL TRIAL: NCT01559753
Title: Comparison of Two Lengths of Treatment in Early-onset Ventilated Associated Pneumonia
Brief Title: Early-onset Ventilator-associated Pneumonia in Adults: Comparison of 8 Versus 15 Days of Antibiotic Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: French Society for Intensive Care (Other); SmithKline Beecham (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHUB/GC001
Record Dates: First submitted 2011-11-29; First posted 2012-03-21 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Pneumonia Ventilator Associated
Keywords: Antibiotic; treatment; ventilator associated pneumonia; duration
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Amoxicillin-Potassium Clavulanate Combination; Ceftriaxone; Cefotaxime; Netilmicin; Tobramycin; Amoxicillin; Clavulanic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 8 days of antibiotic treatment (Experimental): Patients will receive a combination antibiotic during 5 days and then 3 days of a single Beta Lactam antibiotic
  Interventions: Drug: Augmentin, Ceftriaxone, Cefotaxime, netilmycin, tobramycin; Drug: compare 8 to15 days of antibiotic treatment
- 15 days antibiotic treatment (Active Comparator): All patients included in the study will be treated by a combination of antibiotics during the first 5 days, then by monotherapy for 10 days according to the group. The beta-lactam antibiotics will be administered in high doses during the first 3 days of treatment. Aminoglycosides will be administered in a single daily dose, with a loading dose the first day of treatment.
  Interventions: Drug: compare 8 to15 days of antibiotic treatment

INTERVENTIONS:
Drug: Augmentin, Ceftriaxone, Cefotaxime, netilmycin, tobramycin — All patients included in the study will be treated by a combination of antibiotics during the first 5 days, then by monotherapy for either 3 or 10 days according to their allocated group.
  * Beta-Lactams:
    * Amoxicillin + clavulanic Acid : 2 g TDS for 3 days, then 1 g TDS
    * Ceftriaxone : 2 g OD during 3 days, then 1 g OD
    * Cefotaxime : 2 g TDS during 3 days, then 1 g TDS
  * Aminoglycosides
    * Tobramycin : loading dose of 6 mg/kg OD, then 5 mg/kg OD (adaptation in case of renal failure)
    * Netilmicin : loading dose of 10 mg/kg OD, then 8 mg/kg OD (adaptation in case of renal failure)
    * Dibekacin : loading dose of 6 mg/kg OD, then 5 mg/kg OD (adaptation in case of renal failure)
  Other Names: Amoxicillin; Clavulanic acid
  Arms: 8 days of antibiotic treatment
Drug: compare 8 to15 days of antibiotic treatment — All patients included in the study will be treated by a combination of antibiotics during the first 5 days, then by monotherapy for either 3 or 10 days according to their allocated group.
  •
  Beta-Lactams:
  * Amoxicillin + clavulanic Acid : 2 g TDS for 3 days, then 1 g TDS
  * Ceftriaxone : 2 g OD during 3 days, then 1 g OD
  * Cefotaxime : 2 g TDS during 3 days, then 1 g TDS
  Aminoglycosides
  * Tobramycin : loading dose of 6 mg/kg OD, then 5 mg/kg OD (adaptation in case of renal failure)
  * Netilmicin : loading dose of 10 mg/kg OD, then 8 mg/kg OD (adaptation in case of renal failure)
  * Dibekacin : loading dose of 6 mg/kg OD, then 5 mg/kg OD (adaptation in case of renal failure)
  Other Names: Amoxicillin; Clavulanic acid

SUMMARY:
The duration of treatment of community acquired pulmonary infection varies between 5 and 14 days according to the authors (22), or even 3 days with new drugs having long half-life (2). For nosocomial pulmonary infection, treatment durations are not standardized (5). It is simply mentioned the concept of "usual" treatment of at least 15 days. However, recent studies used 10 days of treatment without significant decrease in the rate of healing compared to usual treatment. It is essential to clarify the optimal duration of antibiotic treatment. Indeed, any excessive extension of treatment may increase the occurrence of adverse effects (renal toxicities, hepatic...), and induce resistance of bacteria to antibiotics (selection pressure), colonization of the patient by Multiresistant bacteria and an increase in the cost of treatment

DETAILED DESCRIPTION:
This is a prospective, randomized, open, multi-center study.

3.1 Primary Objective

Show that antibiotic therapy of 8 or 15 days is equivalent in terms of clinical cure rates in the treatment of early onset nosocomial pulmonary infection in patients under mechanical ventilation.

3.2 Secondary Objective

* Study of nosocomial infections: assessing the influence of the duration of antibiotic treatment on the rate of fatal pulmonary and extra-pulmonary infection (definition of nosocomial infections: annex XIII).

  • Study of bacterial Ecology: research of changes in the flora of the gut under treatment and analysis of pathological samples (antibiotic resistance phenotypes +/-genotypes).
* Economic Survey: analyze the costs related to the treatment of nosocomial pneumonia and its complications in two study groups.

ELIGIBILITY:
Inclusion Criteria:

Early onset nosocomial pneumonia in patients under mechanical ventilation since at least 24 h Patients aged 18 years or more The patient must be able to receive either one of the two arms of treatment defined for the study Information on the patient and his family informed consent obtained during the first three days Bacteria sensitive to the specified antibiotic regimen

Exclusion Criteria:

* Patients do not match the criteria for inclusion
* 18 years of age, pregnant Patients
* Another infectious outbreak documented the day of the BAL.
* Patients with acquired immunosuppression (blood diseases, HIV,...), induced (immunosuppressive drugs, cancer, radiation therapy) or congenital.
* Steroids for a period exceeding 15 days.
* Leukopenia (1000 GB/mm (or neutropenia (500 PN/mm)
* Purulent pleural effusion, pulmonary abscess
* Cystic fibrosis
* Antibiotic treatment according to the following terms:

  1. Ongoing curative antibiotic therapy
  2. Antibiotics within 3 days before the diagnosis of VAP, except surgical antibiotic prophylaxis (defined according to the consensus conference "antibiotic prophylaxis in the surgical environment in adult" December 11, 1992) (27)
  3. Use of antibiotics not authorized in the study (see list)
* Allergy to antibiotics used in the study
* Inclusion in another study assessing antibiotic treatment, either the treatment or prevention of nosocomial pulmonary disease
* Refusal to participate
* Lack of informed consent by the patient or his family

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 1998-01; Primary Completion 2002-09 (Actual); Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Cure of respiratory infection | 21 days after inclusion
  The primary endpoint of the present study was the clinical cure rate at day 21. Complete clinical recovery was determined by the absence of the following criteria: death, septic shock (except when associated with a documented non-respiratory infection), intercurrent adverse event attributable to the protocol (or for which attributability to the protocol could not be ruled out) requiring modified antibiotic treatment, and patients who relapsed.

SECONDARY OUTCOMES:
Rate of secondary infections | 21 days
  The study focused on establishing incidence of secondary nosocomial infections; number of patients on antibiotic treatment; total number of days of antibiotic treatment; duration of MV; number of patients still under ventilation; number of patients still in ICU; length of stay in ICU on day 21; and mortality rate at 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles R CAPELLIER, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Besancon

REFERENCES:
- [Derived] Capellier G, Mockly H, Charpentier C, Annane D, Blasco G, Desmettre T, Roch A, Faisy C, Cousson J, Limat S, Mercier M, Papazian L. Early-onset ventilator-associated pneumonia in adults randomized clinical trial: comparison of 8 versus 15 days of antibiotic treatment. PLoS One. 2012;7(8):e41290. doi: 10.1371/journal.pone.0041290. Epub 2012 Aug 31. PMID 22952580